CLINICAL TRIAL: NCT05681091
Title: The Effect of Perioperative Hypothermia on Postoperative Pain and Pain Sensitization With Laparoscopic Surgery: a Prospective Observational Study
Brief Title: Effect of Perioperative Hypothermia on Postoperative Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Body temperature and pain
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to observe the impact of perioperative body temperature on postoperative pain and pain sensitization for the patients with laparoscopic surgery. Based on this study the investigators aimed to explore the effect of perioperative hypothermia on postoperative pain.

DETAILED DESCRIPTION:
This study aims to included surgery patients to observe the impact of perioperative body temperature on postoperative pain and pain sensitization for the patients with laparoscopic surgery. Body temperature and postoperative pain will be continuously assessed, and then association analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old
* American society of anesthesiologists I-III
* Patients who plan to laparoscopic surgery under general anesthesia
* Volunteer to participate in this study and sign informed consent.

Exclusion Criteria:

* the patient with chronic pain
* Patients with fever
* The patient is infected
* Severe vision, hearing, language impairment or other reasons unable to communicate with visitors
* Patients with known mental illness or lack of communication or cognitive impairment before operation;
* Long-term use of sedatives, antidepressants or alcoholism
* Artificial cooling and low temperature protection were taken during the operation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the patients' age is during 18-70 years old
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Patients' pain score after surgery | From ending of the surgery to 24 hours after anesthetic resuscitation
  The patients' pain score was tested with Numerical analogue scale of pain (0-10, 0 represents pain free, and 10 represents unbearable pain).

SECONDARY OUTCOMES:
Patients' pain score during postanesthesia care unit | From ending of the surgery to the time when discharge from postanesthesia care unit with a mean of 30 minutes after surgery
  The patients' pain score was tested with Numerical analogue scale of pain (0-10, 0 represents pain free, and 10 represents unbearable pain).
Pressure pain threshold | From beginning of the surgery to the time when discharge from postanesthesia care unit with a mean of 30 minutes after surgery
  the patients' pain threshold was tested by tenderness meter.

CONTACTS AND LOCATIONS:
Overall Officials: Huang He, MD, Study Director — Department of Anesthesiology, The Second Affiliated Hospital, Chongqing
Locations (1):
- Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China